CLINICAL TRIAL: NCT04927507
Title: Rotator Cuff Injury Managed With ERAS and Internet Plus Nursing
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Second Affiliated Hospital, School of Medicine, Zhejiang University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2021-0061
Record Dates: First submitted 2021-06-03; First posted 2021-06-16 (Actual); Last update posted 2021-06-16 (Actual); Status verified 2021-06

CONDITIONS: Rotator Cuff Injuries
MeSH Terms: conditions — Rotator Cuff Injuries

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control group (No Intervention): The control group was given routine nursing.
- Observation group (Experimental): The observation group was given the Internet plus nursing home rehabilitation mode.
  Interventions: Behavioral: Internet plus nursing home rehabilitation

INTERVENTIONS:
Behavioral: Internet plus nursing home rehabilitation — The observation group was given the Internet plus nursing home rehabilitation mode.
  Relying on mobile app and wechat public service platform, patients can get online guidance of rehabilitation training video through app and wechat, and get professional rehabilitation guidance at any time.
  Arms: Observation group

SUMMARY:
Rotator cuff injury patients treated with ERAS were included. The control group was given routine nursing. The observation group was given the Internet plus nursing home rehabilitation mode.

Relying on mobile app and wechat, patients can get online guidance of rehabilitation training video through app and wechat, and get professional rehabilitation guidance at any time.

ELIGIBILITY:
Inclusion Criteria:

* Rotator cuff injury
* ERAS surgery treatment
* Full thickness tear of rotator cuff, The range of tear is 1cm-3cm

Exclusion Criteria:

* Surgery not applicable
* Combined with other injuries, malignant tumor, disabilities, mental illness, critically ill patients, pregnant women, illiteracy, minors, cognitive impairment

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 140 (Estimated)
Dates: Start 2020-01-01 (Actual); Primary Completion 2021-12-31 (Estimated); Study Completion 2022-12-31 (Estimated)

PRIMARY OUTCOMES:
The Constant-Murley score | up to 6 months
  The Constant-Murley score (CMS) is a 100-points scale composed of a number of individual parameters. These parameters define the level of pain and the ability to carry out the normal daily activities of the patient. The Constant-Murley score was introduced to determine the functionality after the treatment of a shoulder injury. The best situation is 100 points. The worst situation is 0 points.

CONTACTS AND LOCATIONS:
Locations (1):
- Ping Qian, Hangzhou, China

IPD SHARING:
Plan to Share IPD: No